CLINICAL TRIAL: NCT03900585
Title: Physical Activity and Fatigue in Danish Patients With Myasthenia Gravis - an Intervention Study
Brief Title: Can Interval Walking Influence on Fatigue in the Danish Cohort of Myasthenia Gravis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restricted and new rules for data protection, the use of an app could not be approved
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Linda Kahr Andersen, Master of Health Science, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18031231
Record Dates: First submitted 2019-02-25; First posted 2019-04-03 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval walking (Experimental): Interval walking for 10 weeks, 150 minutes per week administered by an app on the patient's telephone.
  Interventions: Behavioral: Interval walking
- Control (No Intervention): Patients live as normal, though aerobe training restricted to a maximum of 30 minutes a week.

INTERVENTIONS:
Behavioral: Interval walking — Interval walking administered by an app on the patient's telephone. Interval walking for 150 minutes/week for 10 weeks.
  Arms: Interval walking

SUMMARY:
The study is a controlled, randomized intervention trial. Patients are randomized into either an intervention group or a control group. The duration of the study is 10 weeks. Patients in the intervention group participate in a 10 weeks exercise program consisting of 150 minutes interval walking per week administered by an app on the patient's telephone. Patients in the control group live as usually, with a maximum of 30 minutes aerobic exercise per week.

Before and after the 10 weeks study period, patients (from both the intervention and the control group) participate in a 2 hours session of functional testing (e.g. walk tests, test of muscle strength ect.) at Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed informed consent.
* Able to read and understand Danish or English.
* Diagnosed with mild to moderate myasthenia gravis (I-IV on the Myasthenia Gravis Foundation of American Clinical Classification, MGFA).
* Documented history of acetylcholine receptor (AChR) or Muscle Specific Kinase (MuSK) antibody positive, or abnormal repetitive nerve stimulation testing (decrement > 10%) on EMG or abnormal single fiber EMG (conduction block or jitter) or based on their clinical history and symptom improvement with acethylcholinesterase inhibitors.
* If the patient is on oral corticosteroids, the dose must be stable for at least 1 month prior to inclusion.
* If the patient is on cholinesterase inhibitors the dose must be stable 2 weeks prior to inclusion.

Exclusion Criteria:

* MGFA grade V disease
* Other disorders that are not related to MG, or drugs, that interfere with muscle strength, balance and fatigue.
* Serious medical illness (e.g. uncontrolled insulin dependent diabetes mellitus, symptomatic coronary artery disease, and cancer).
* Dementia or pregnancy.
* Unspecified reasons judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | 6 minutes
  Walk test

SECONDARY OUTCOMES:
30-s sit to stand test | 30 seconds
  How many times in 30 seconds can the patient stand up from sitting on a chair?
Quantitative Myasthenia Gravis Score | 45 minutes
  The Quantitative Myasthenia Gravis (QMG) score is an established and validated measure of disease severity used in myasthenia gravis (MG) trials. This scoring system is based on quantitative testing of sentinel muscle groups by means of a 4 point scale ranging from 0 (no symptoms) to 3 (severe symptoms). The scale measures ocular, bulbar, respiratory and limb function, grading each finding, and the total score ranges from 0(no myasthenic findings) to 39 (maximal myasthenic deficits).
Myasthenia gravis composite score | 30 minutes
  The Myasthenia Gravis composite score (MGC) covers 10 important functional domains most frequently involved in patients with MG. This scoring system is based on quantitative testing of muscle groups, or symptom history told by the patient, by means of a 4 point scale ranging from 0 (no symptoms) to 9 (severe symptoms). The scale measures ocular, bulbar, respiratory and limb function, grading each finding, and the total score ranges from 0(no myasthenic findings) to 50 (maximal myasthenic deficits).
Myasthenia gravis activity of daily living profile (MG-ADL) | 10 minutes
  Impact on daily living is assessed using the MG-ADL. An eight-question survey of symptoms severity, with each response graded from 0 (normal) to 3 (most severe). Questions include ocular, oropharyngeal, respiratory, and extremity functions. Total MG-ADL score ranges from 0 to 24. MG-ADL is also an indirect measurement of disease severity.
Myasthenia gravis quality of life 15-item score (MG-QoL15) | 3 minutes
  MG -specific quality-of-life instrument is a 15-item questionnaire encompassing physical and psychological domains of MG to assess disease-specific Qol in MG patients. Rating consist of a 5-point scale ranging from 0 ("not at all") to 4 ("very much") as to the degree to which patients agree with the given statement summing up to a total score 0-60 points.
Multidimensional Fatigue Inventory (MFI-20) | 5 minutes
  Self-reported questionnaire that measure fatigue severity. It contains 20 items and consists of five domains: mental fatigue, reduced motivation, reduced activity, physical fatigue and general fatigue. The response options consist of five check boxes ranging from "yes, that is true" to "No, that is not true". The scores in each domain range from 4 to 20, with higher scores indicating higher levels of fatigue. A total fatigue score for all five domains is not used. MFI-20 has been used in several clinical and healthe populations.

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, Professor, Study Director — Rigshospitalet, Denmark